CLINICAL TRIAL: NCT01346605
Title: Registry for CARDIAC PERFUSION CT
Acronym: RECRUIT
Status: Withdrawn | Type: Observational
Why Stopped: No funding
Sponsor: MDDX LLC (Industry)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: RECRUIT Study
Record Dates: First submitted 2011-04-30; First posted 2011-05-03 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Coronary Artery Disease
Keywords: Cardiac CT, heart disease
MeSH Terms: conditions — Coronary Artery Disease; Heart Diseases

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CCTA patients: Prior stress SPECT with intermediate to high likelihood to be referred to the cardiac catheterization laboratory for an invasive coronary angiogram or patients presenting with chest pain and clinical indication of Coronary CT Angiography and an initial calcium score above 300

SUMMARY:
This protocol describes a study whose goal is to collect de-identified Cardiac CT Perfusion (CTP) acquisition parameters and clinical findings from approximately 20 qualified medical facilities. The study uses an electronic data capture tool to collect the de-identified data to create a global multi-center registry. This registry will be used for scientific analysis and publication of pertinent medical trends such as CT utilization, radiation dose, and common cardiovascular findings.

DETAILED DESCRIPTION:
The recently developed technique of Cardiac CT Perfusion (CTP) gathers information on both coronary anatomy and myocardial perfusion in a single scan. This diagnostic test can detect the presence of coronary plaque as well as assess the functional significance of a stenosis. To date, it is estimated that 1000 cases of CTP have been performed in the world. While no exceptional adverse events have been reported (nor are expected), the image quality and clinical validation in a multi-center multi-vendor setting has been a marked issue for many experts in this nascent field. This issue has hampered the clinical utility of this test and raises concerns about its widespread utilization leading to unnecessary costs and exposure to radiation.

Historically, the rapid explosion in the use of a related procedure, Cardiac CT Angiography (CCTA) started in 2004 and was marked by large-scale variation in radiation dose, quality issues, inappropriate use, and interpretation proficiency. Critics of the rapid growth of CCTA defamed the procedure for imaging abuse charges and noted unchecked and irresponsible use radiation.

The purpose of RECRUIT is to prevent this clinical inefficiency from occurring again. The main goal of RECRUIT is to determine the best practices for optimal acquisition and interpretation of the CTP images, in an effort to optimize standards before the inevitable rapid adoption of this potentially revolutionary technology. RECRUIT will aim to maximize the clinical effectiveness and minimize the clinical risks associated with CTP before the protocol becomes integrated into the standard-of-care and harmonization of the best practices is nearly impossible.

RECRUIT will enable select clinics that are currently performing CCTA to perform CTP by training them on the latest acquisition techniques as provided by the field leaders in CTP. In addition to providing the acquisition protocol, our researchers will provide the clinical team with a sophisticated EDC tool that effectively monitors numerous factors that could influence the quality of the images. Finally, RECRUIT will collect de-identified images from the sites for analysis in our core lab. Analysis of the images will be correlated with acquisition techniques and patient factors (i.e. BMI). This information fed back to the clinical team that performed the procedure in an effort to improve their proficiency. This process will proceed in an iterative manner, with all endpoints being tracked for reporting in peer-reviewed literature.

ELIGIBILITY:
Inclusion Criteria:

* Moderate-high likelihood of coronary artery disease with a prior stress SPECTMPI exam likely to be referred to the cardiac catheterization laboratory for invasive angiogram or patients presenting with clinical indication of Coronary -CT Angiography and an initial calcium score above 300
* Stable angina or anginal equivalent as the chief symptom.
* Age > 34 years old
* Able to comprehend and sign the consent form.

Exclusion Criteria:

* BMI<41
* Acute coronary syndromes (unstable angina, non-ST elevation myocardial infarction, ST elevation myocardial infarction)
* Unstable clinical conditions (i.e. hemodynamic instability, arrhythmias)
* Premenopausal women who have menstruated in the last year
* Glomerular Filtration Rate (GFR) < 60 ml/min/BSA as an indicator of renal insufficiency
* Known allergy to iodinated contrast agents
* Patients who are on metformin medication for any reason
* Atrial fibrillation
* Asthma
* Critical aortic stenosis
* Systolic blood pressure < 90 mmHg
* Advanced heart block
* Pacemaker or AICD

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prior stress SPECT with intermediate to high likelihood to be referred to the cardiac catheterization laboratory for an invasive coronary angiogram or patients presenting with chest pain and clinical indication of Coronary CT Angiography and an initial calcium score above 300
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Best Practices for CTP | 2 years
  Collect DICOM cases and determine the best practices for CTP, including radiation dose, image quality and patient comfort

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Cury, MD, Principal Investigator — Miami Baptist; James Min, MD, Study Chair — Cedars Sinai
Locations (1):
- Miami Baptist, Miami, Florida, United States